CLINICAL TRIAL: NCT06628869
Title: The Effects of Oral Fructanase Administration on Gastrointestinal Symptoms After Inulin Challenge in Healthy Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BIO-CAT, Inc. (Industry)
Collaborators: Biofortis, Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: BCCT-AMS-0011; BIO-2407 (Other: Biofortis, Inc.)
Record Dates: First submitted 2024-10-03; First posted 2024-10-08 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Digestive Health; Gastrointestinal Health; FODMAP Intolerance; Food Sensitivity
Keywords: digestive enzyme; FODMAP; fructanase; inulinase; fructan hydrolyase; enzyme; food sensitivity; inulin; bloating; flatulence; fermentation; methane; hydrogen; dietary supplement; dietary fiber; food intolerance; fructan; oligosaccharide; fructooligosaccharide; inulinooligosaccharide; fructo-oligosaccharide; inulino-oligosaccharide; non-starch polysaccharidase; NSPase; carbohydrate-active enzyme; CAZyme; microbiome; metagenome; food challenge
MeSH Terms: conditions — Food Intolerance; Flatulence | interventions — levanase; inulinase; beta-Fructofuranosidase

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fructanase (Active Comparator): Total 400 inulinase activity units (INU) per dose
  Interventions: Dietary Supplement: Fructanase
- Placebo (Placebo Comparator): Maltodextrin
  Interventions: Dietary Supplement: Maltodextrin placebo

INTERVENTIONS:
Dietary Supplement: Fructanase — Participants will consume one capsule containing 400 INU inulinase (325 mg, includes maltodextrin) with a mixture of oatmeal (40 grams) and inulin (25 grams). Participants will be directed to consume the capsule after two spoonfuls of oatmeal. The fructanase was obtained from Aspergillus tubingensis.
  Other Names: inulinase; fructan hydrolase; beta-fructofuranosidase; beta-fructosidase
  Arms: Fructanase
Dietary Supplement: Maltodextrin placebo — Participants will consume one capsule containing 300 mg maltodextrin with a mixture of oatmeal (40 grams) and inulin (25 grams). Participants will be directed to consume the capsule after two spoonfuls of oatmeal. The maltodextrin was obtained from tapioca.
  Arms: Placebo

SUMMARY:
The carbohydrate inulin (from chicory root) is a healthy prebiotic ingredient found in dietary supplements and fortified foods (Nagy et al). Inulin is representative of a broader class of typically health-associated, yet fermentable carbohydrates called fructans that occur naturally in many vegetables, fruits, and wheat. Fructans, or long chains of fructose units, are resistant to human digestive enzyme hydrolysis and transit intact to the small intestine and colon where they undergo rapid fermentation by intestinal microbes. This microbial metabolism of fructans produces gas and other fermentation byproducts that can lead to excess gastrointestinal (GI) symptoms like abdominal bloating, cramping, stomach rumbling, and flatulence (Bonnema et al; Briet et al; Bruhwyler et al), especially in individuals with irritable bowel syndrome (Van den Houte et al). A new digestive enzyme called fructanase was developed to help with GI symptoms associated with fructan consumption. Positive findings from in vitro digestion simulations (Guice et al) and a first-in-human safety trial (Garvey et al) helped define the fructanase dose for this clinical trial-the primary objective of which is to investigate the effect of oral fructanase administration on GI symptoms in healthy adults after consuming oatmeal with added inulin (25 grams). Secondary outcomes include breath hydrogen and methane levels, which serve as biomarkers of intestinal microbial fermentation. The investigators hypothesize that fructanase administration will lower the severity of GI symptoms after inulin consumption, as well as lower breath biomarkers of intestinal microbial fermentation, compared to placebo.

DETAILED DESCRIPTION:
Fructanase (also known as inulinase, fructan hydrolase, beta-fructosidase, and beta-fructofuranosidase) represents an innovative enzymatic approach to hydrolyze dietary fructans and improve fructan-type fermentable oligo-, di-, monosaccharides, and polyols (FODMAP) tolerance. We have previously shown in vitro that a microbial fructanase (obtained by fermentation of Aspergillus tubingensis) effectively hydrolyzes a variety of dietary inulins and fructans following simulated oro-gastric digestion in the static INFOGEST model [Guice et al]. We have also completed a Phase I clinical trial in healthy adults demonstrating the safety and tolerability of twice daily fructanase supplementation (total 2,000 inulinase activity units (INU) per day) for 4 weeks [Garvey et al]. Despite its safety and promising application in nutrition and GI health, rigorous clinical evaluation of fructanase's efficacy in improving GI tolerance to fructans is warranted.

This is a randomized, double-blind, two-period crossover study with one screening visit (Visit 1, Day -7) and two test visits (Visits 2 and 3; Days 0 and 7). Participants will arrive for their screening visit on Day -7. After participants provide voluntary informed consent, participants will undergo medical history, prior and current medication/supplement use, inclusion and exclusion criteria assessments, and last menses query (if applicable). Additionally, height, body weight, and vital signs will be measured, and theoretical body mass index (BMI) will be calculated. An in-clinic urine pregnancy test will be performed on all female participants. Participants will be instructed to maintain physical activity and habitual diet as much as possible while abstaining from supplements, beverages, or food products with digestive enzymes, prebiotic ingredients, live probiotics (e.g., yogurt, kombucha), or postbiotic ingredients prior to Visit 2 (Day 0). Those who are taking exclusionary supplements, foods, and beverages will be instructed to stop taking these products, and their Visit 2 (Day 0) will be scheduled to allow for the appropriate pre-randomization washout period. Additionally, pre-menopausal female participants will be scheduled to allow their Visit 2 (Day 0) to occur during the menstrual cycle follicular phase (defined as days 1-14 of the menstrual cycle, with day 1 as the first day of menses). To all participants, a standardized low FODMAP meal will be dispensed with instructions to consume the meal in its entirety the evening prior to Visit 2 (Day 0). The instructions will include timing of meal consumption in order to maintain the appropriate fast. Participants will also be instructed to follow a low FODMAP diet the day prior to Visit 2, while also being reminded to abstain from alcohol consumption for 48 h, to abstain from vigorous exercise for 24 h, to fast (≥10 h; water only), and to brush their teeth in the morning prior to Visit 2 (Day 0).

At Visit 2 (Day 0), participants will arrive at the clinic in a fasting state (≥10 h; water only). Eligible participants will undergo clinic visit procedures (concomitant medication/supplement use, assess inclusion/exclusion criteria, and body weight), last menses query (where applicable), and adverse event (AE) assessment. Participants will be queried about compliance with study instructions and changes to habitual lifestyle, diet, and alcohol consumption. At t = -0.25 h (± 5 min), where t = 0 h is the time of study product consumption, participants will provide a breath sample for hydrogen and methane analysis and complete a questionnaire to assess baseline GI symptoms prior to study product consumption. Participants will then be randomized to a study product sequence and will be administered their assigned study product capsule (fructanase or placebo) that will be consumed with oatmeal and 25 g of inulin (t = 0 h). In addition, 8 oz. of water will be provided. Participants will be allowed up to 10 minutes to completely consume the oatmeal and inulin mixture, with fructanase or placebo, with t = 0 h designated as the start of study product consumption. Following study product consumption, participants will complete the GI symptom questionnaire and provide a breath sample for hydrogen and methane analysis at t = 1, 2, 3, 4, 5, 6, 7, and 8 h (± 5 min). Participants will also be provided with 8 oz. of water at t = 2 and 4 h. Participants will be allowed to drink each 8 oz. of water ad libitum over each 2 h period, but the entire 8 oz. of water must be consumed prior to the next water administration (e.g., drink all 8 oz. provided at t = 2 h prior to the next water administration at t = 4 h). A standard low FODMAP lunch with 8 oz. of water will be provided after the t = 6 h assessments.

Prior to departure from the study center, AEs will be assessed, then study instructions will be provided, including: 1) maintaining habitual physical activity, 2) continuing to follow the low FODMAP diet for the remainder of the day, 3) abstaining from alcohol consumption for the remainder of the day, and 4) abstaining from supplements, beverages, or food products with digestive enzymes, prebiotic ingredients, live probiotics (e.g., yogurt, kombucha), or postbiotic ingredients throughout the study. The same standardized low FODMAP meal consumed the evening prior to Visit 2 will be dispensed with instructions to consume the meal in its entirety the evening prior to Visit 3 (Day 7). The instructions will include timing of meal consumption in order to maintain the appropriate fast. Participants will also be instructed to follow a low FODMAP diet the day prior to Visit 3 (Day 7), while also being reminded to abstain from alcohol consumption for 48 h, to abstain from vigorous exercise for 24 h, to fast (≥10 h; water only), and to brush their teeth in the morning prior to Visit 3 (Day 7).

The following morning (Day 1), participants will receive an email link at t = 24 h to complete a series of brief questionnaires, including:

* Modified Single-Item Sleep Quality Scale
* Single-Item Stool Consistency Scale
* GI-VAS assessing symptoms "since participant left the clinic"
* A single question to confirm compliance with study instructions.

Participants will be instructed to complete these questionnaires the morning of Day 1 after their first bowel movement or immediately prior to their usual lunch time, whichever occurs first.

At Visit 3 (Day 7), participants will arrive at the clinic fasted (≥10 h; water only) and undergo clinic visit procedures, including: concomitant medication/supplement use, review inclusion/exclusion criteria, and body weight, last menses query (if applicable), and AE assessment. Participants will be queried about compliance with study instructions and changes to habitual lifestyle, diet, and alcohol consumption. Participants will then complete all study procedures outlined in Visit 2 (except for randomization). The same timing and volume of water consumed at Visit 2 will be replicated at Visit 3. The same lunch (items and quantity) consumed at Visit 2 will be replicated at Visit 3.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, age ≥20 to ≤50 y at Visit 1 (Day -7).
2. BMI ≥18.5 to less than 30.0 kg/m2 at Visit 1 (Day -7).
3. Non-user (never used, or former user defined as cessation ≥12 months) of tobacco or nicotine products (e.g., cigarette smoking, vaping, chewing tobacco) with no plans to begin use during the study period.
4. Willing to maintain habitual diet, physical activity, and body weight throughout the trial.
5. Willing to refrain from exclusionary medications, supplements, and products throughout the study.
6. No health conditions that would prevent him/her from fulfilling the study requirements as judged by the Clinical Investigator on the basis of medical history and routine laboratory test results.
7. Understands the study procedures and signs forms providing informed consent to participate in the study and authorizes the release of relevant protected health information to the Clinical Investigator.

Exclusion Criteria:

1. Known sensitivity, intolerability, or allergy to any of the study products or their excipients.
2. Clinically important GI condition that would potentially interfere with the evaluation of the study product (e.g., inflammatory bowel disease, irritable bowel syndrome, gastroesophageal reflux disease requiring any medication, dyspepsia, Crohn's disease, celiac disease, history of surgery for weight loss, gastroparesis, and clinically significant lactose or gluten intolerance or other food or ingredient allergies).
3. Recent (within 2 weeks of Visit 1; Day -7) history of an episode of acute GI illness such as nausea/vomiting or diarrhea (defined as ≥3 loose or liquid stools/d).
4. Self-reported history (within 6 weeks of Visit 1; Day -7) of constipation (defined as fewer than 3 bowel movements per week).
5. Uncontrolled and/or clinically important pulmonary (including uncontrolled asthma), cardiac (including, but not limited to, atherosclerotic disease, history of myocardial infarction, peripheral arterial disease, stroke), hepatic, renal, endocrine (including Type 1 and Type 2 diabetes mellitus), hematologic, immunologic, neurologic (such as Alzheimer's or Parkinson's disease), psychiatric (including depression and/or anxiety disorders) or biliary disorders. Conditions which are well-controlled or resolved will be assessed by the Clinical Investigator on a case-by-case basis.
6. Uncontrolled hypertension (systolic blood pressure ≥140 mm Hg or diastolic blood pressure ≥90 mm Hg) as defined by the blood pressure measured at Visit 1 (Day -7). Stable use of hypertension medication is allowed [defined as no change in medication regimen within the 3 months prior to Visit 1 (Day -7)].
7. Have received a COVID-19 vaccine within 2 weeks of randomization or expected to receive a COVID-19 vaccine during the study period.
8. Had a positive SARS-CoV2 test and experienced symptoms for more than 2 months (i.e. "long-haulers").
9. Extreme dietary habits (e.g., vegetarian, vegan, Atkins diet, etc.) at the discretion of the Clinical Investigator.
10. History or presence of cancer in the prior 2 years, except for non-melanoma skin cancer.
11. Major trauma or any other surgical event within 3 months of Visit 1 (Day -7).
12. Signs or symptoms of an active infection of clinical relevance within 5 days of Visit 1 (Day -7). The visit may be rescheduled such that all signs and symptoms have resolved (at the discretion of the Clinical Investigator) at least 5 days prior to Visit 1 (Day -7).
13. Weight loss or gain more than 4.5 kg in the 3 months prior to Visit 1 (Day -7).
14. Currently or planning to be on a weight loss regimen during the study.
15. Use of weight loss medications, incretin mimetics, and/or GLP-1 agonists in the 3 months prior to Visit 1 (Day -7).
16. Consumption of supplemental inulin/chicory root or inulin/chicory root-fortified foods and beverages equivalent to more than 10 g inulin per day within 1 month of Visit 1 (Day -7).
17. Antibiotic use within 3 months of Visit 1 (Day -7) and throughout the study period.
18. Use of steroids within 1 month of Visit 1 (Day -7) and throughout the study period.
19. Habitual use (i.e., daily) of marijuana and hemp products including CBD products within 30 days of Visit 1 (Day -7).
20. Chronic use (i.e., daily on a regular basis) of anti-inflammatory medications (e.g., NSAIDS) within 1 month of Visit 1 (Day -7).
21. Use of medications (over-the-counter or prescription) and/or dietary supplements, known to influence GI function, including but not limited to, digestive enzymes, pre- and probiotic supplements as well as foods or beverages containing live probiotics (e.g., yogurt, kombucha), fiber supplements, laxatives, enemas, suppositories, H2 blockers, proton pump inhibitors, antacids, anti-diarrheal agents, anti-depressants, and/or anti-spasmodics within 2 weeks of Visit 1 (Day -7) and throughout the study period. Standard multivitamin and mineral supplements are allowed.
22. Participated in endoscopy or endoscopy preparation within 3 months prior to Visit 1 (Day -7).
23. Exposure to any non-registered drug product within 4 weeks prior to Visit 1 (Day -7).
24. Female who is pregnant, planning to be pregnant during the study period, lactating, or is of childbearing potential and is unwilling to commit to the use of a medically approved form of contraception throughout the study period. Participants who are pregnant during the study will be discontinued.
25. Recent history (within 12 months of screening; Visit 1; Day -7) of alcohol or substance abuse. Alcohol abuse is defined as more than 14 drinks per week (1 drink = 12 oz beer, 5 oz wine, or 1½ oz distilled spirits).
26. Receipt or use of study products in another research study within 4 weeks prior to Visit 2 (Day 0) or longer if the previous study product is deemed by the Clinical Investigator to have lasting effects that might influence the eligibility criteria or outcomes of current study.
27. Has a condition the Clinical Investigator believes would interfere with the participant's ability to provide informed consent, comply with the study protocol, which might confound the interpretation of the study results, or put the participant at undue risk.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2024-11-04 (Actual); Primary Completion 2024-12-16 (Actual); Study Completion 2024-12-17 (Actual)

PRIMARY OUTCOMES:
Maximum postprandial baseline-adjusted overall abdominal symptoms severity over the 8-hour in-clinic period | 8 hours
  The primary endpoint is the difference in the maximum postprandial baseline-adjusted overall abdominal symptoms visual analog scale (VAS) score over the 8-hour in-clinic period between placebo and fructanase treatments. Participants will rate overall abdominal symptoms severity from "excellent, none at all" (score: 0) to "really awful, the worst it has been" (score: 100). Participants will be instructed to rate themselves by marking the VAS at the point that was most appropriate to their feeling over the prior hour. The distance from the point marked on the VAS to the left end of the scale will be measured in millimeters. The change from baseline is calculated by subtracting the baseline score from the score at each postprandial time point. At Visits 2 and 3 (Days 0 and 7), the VAS will be administered in-clinic at t = -0.25, 1, 2, 3, 4, 5, 6, 7, and 8 hours.

SECONDARY OUTCOMES:
Maximum postprandial unadjusted overall abdominal symptoms severity over the 8-hour in-clinic period | 8 hours
  Difference in the maximum postprandial unadjusted overall abdominal symptoms visual analog scale (VAS) score over the 8-hour in-clinic period between placebo and fructanase treatments. Participants will rate overall abdominal symptoms severity from "excellent, none at all" (score: 0) to "really awful, the worst it has been" (score: 100). Participants will be instructed to rate themselves by marking the VAS at the point that was most appropriate to their feeling over the prior hour. The distance from the point marked on the VAS to the left end of the scale will be measured in millimeters. At Visits 2 and 3 (Days 0 and 7), the VAS will be administered in-clinic at t = -0.25, 1, 2, 3, 4, 5, 6, 7, and 8 hours.
Maximum postprandial baseline-adjusted and unadjusted individual gastrointestinal symptom severity over the 8-hour in-clinic period | 8 hours
  Difference in the maximum postprandial baseline-adjusted and unadjusted gastrointestinal symptom visual analog scale (VAS) score over the 8-hour in-clinic period between placebo and fructanase treatments. Participants will rate gastrointestinal symptom severity from "excellent, none at all" (score: 0) to "really awful, the worst it has been" (score: 100). Participants will be instructed to rate themselves by marking the VAS at the point that was most appropriate to their feeling over the prior hour. The distance from the point marked on the VAS to the left end of the scale will be measured in millimeters. For baseline-adjusted scores, the distance from the point marked on the VAS to the left end of the scale will be measured in millimeters. At Visits 2 and 3 (Days 0 and 7), the VAS will be administered in-clinic at t = -0.25, 1, 2, 3, 4, 5, 6, 7, and 8 hours. Individual symptoms to be queried include abdominal bloating, abdominal pain, flatulence, burping, stomach rumbling, nausea, an
Total gastrointestinal symptom burden over the 8-hour in-clinic period represented by the visual analog scale (VAS) score area-under-the-curve (AUC) and baseline-adjusted positive area-under-the-curve (p-AUC): | 8 hours
  Symptoms to be queried include overall abdominal symptoms, abdominal bloating, abdominal pain, flatulence, burping, stomach rumbling, nausea, and fatigue
Time to maximum gastrointestinal symptom visual analog scale (VAS) score over the 8-hour in-clinic period | 8 hours
  Symptoms to be queried include overall abdominal symptoms, abdominal bloating, abdominal pain, flatulence, burping, stomach rumbling, nausea, and fatigue
Maximum 24-hour gastrointestinal symptom visual analog scale (VAS) score, representing the time since leaving the clinic | 24 hours
  Symptoms to be queried include overall abdominal symptoms, abdominal bloating, abdominal pain, flatulence, burping, stomach rumbling, nausea, and fatigue
Change over time, from 0 to 8 hours, in the gastrointestinal symptom visual analog scale (VAS) score | 8 hours
  Symptoms to be queried include overall abdominal symptoms, abdominal bloating, abdominal pain, flatulence, burping, stomach rumbling, nausea, and fatigue
Change over time, from 0 to 24 hours, in the gastrointestinal symptom visual analog scale (VAS) score | 24 hours
  Symptoms to be queried include overall abdominal symptoms, abdominal bloating, abdominal pain, flatulence, burping, stomach rumbling, nausea, and fatigue
Sleep quality | 24 hours
  The Modified Single-Item Sleep Quality Scale (mSI-SQS) will be completed by each participant electronically (i.e., outside of the clinic visit) after awakening the morning of Days 1 and 8, which will be approximately 24 h (± 1 h) after consuming the assigned study product at Visits 2 and 3 (Days 0 and 7). The SI-SQS has previously been validated as a weekly questionnaire [Snyder et al]. The mSI-SQS directs the participant to rate the overall quality of sleep over the prior night by marking an integer score from 0 to 10, according to the following 5 categories: 0 = terrible, 1-3 = poor, 4-6 = fair, 7-9 = good, and 10 = excellent. When rating their sleep quality, participants are instructed to consider the following core components of sleep quality: how many hours of sleep they had, how easily they fell asleep, how often they woke up during the night (except to go to the bathroom), how often they woke up earlier than they had to in the morning, and how refreshing their sleep was.
Stool consistency | 24 hours
  On the morning of Days 1 and 8, a Single-Item Stool Consistency Scale (SI-SCS) will be used to capture participant reported stool consistency ~24 h following study product consumption. Specifically, participants will rate the consistency of their stool since they left the clinic yesterday compared to their usual stool consistency, with the following options: 0 = Not applicable-no bowel movement occurred; 1 = Significantly more firm (hard) than usual; 2 = Slightly more firm (hard) than usual; 3 = Usual consistency; 4 = Slightly more loose (soft) than usual; 5 = Significantly more loose (soft) than usual.
Breath hydrogen Cmax (ppm) | 8 hours
  Maximum concentration
Breath hydrogen concentration AUC (ppm × min) | 8 hours
  Area-under-the-curve
Breath hydrogen Tmax (min) | 8 hours
  Time to maximum concentration
Breath methane Cmax (ppm) | 8 hours
  Maximum concentration
Breath methane Tmax (min) | 8 hours
  Time to maximum concentration
Breath combined hydrogen and methane Cmax (ppm) | 8 hours
  Maximum concentration
Breath combined hydrogen and methane concentration AUC (ppm × min) | 8 hours
  Area-under-the-curve
Breath combined hydrogen and methane Tmax (min) | 8 hours
  Time to maximum concentration
Breath methane concentration AUC (ppm × min) | 8 hours
  Area-under-the-curve
Exit survey results | 8 days
  The exit survey directed participants to (i) choose their suspected treatment sequence (digestive enzyme first or placebo first), and (ii) select their confidence in selection in choice of suspected treatment sequence assessed using a categorical 5-point Likert scale.

CONTACTS AND LOCATIONS:
Overall Officials: Aditi M. Shaw, MD, Principal Investigator — Biofortis, Inc.
Locations (1):
- Biofortis, Inc., Addison, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Snyder E, Cai B, DeMuro C, Morrison MF, Ball W. A New Single-Item Sleep Quality Scale: Results of Psychometric Evaluation in Patients With Chronic Primary Insomnia and Depression. J Clin Sleep Med. 2018 Nov 15;14(11):1849-1857. doi: 10.5664/jcsm.7478. PMID 30373688
- [Background] Garvey SM, LeMoire A, Wang J, Lin L, Sharif B, Bier A, Boyd RC, Baisley J. Safety and Tolerability of Microbial Inulinase Supplementation in Healthy Adults: A Randomized, Placebo-Controlled Trial. Gastro Hep Adv. 2024 Jun 21;3(7):920-930. doi: 10.1016/j.gastha.2024.05.013. eCollection 2024. PMID 39318719
- [Background] Briet F, Achour L, Flourie B, Beaugerie L, Pellier P, Franchisseur C, Bornet F, Rambaud JC. Symptomatic response to varying levels of fructo-oligosaccharides consumed occasionally or regularly. Eur J Clin Nutr. 1995 Jul;49(7):501-7. PMID 7588500
- [Background] Bruhwyler J, Carreer F, Demanet E, Jacobs H. Digestive tolerance of inulin-type fructans: a double-blind, placebo-controlled, cross-over, dose-ranging, randomized study in healthy volunteers. Int J Food Sci Nutr. 2009 Mar;60(2):165-75. doi: 10.1080/09637480701625697. PMID 18608562
- [Background] Bonnema AL, Kolberg LW, Thomas W, Slavin JL. Gastrointestinal tolerance of chicory inulin products. J Am Diet Assoc. 2010 Jun;110(6):865-8. doi: 10.1016/j.jada.2010.03.025. PMID 20497775
- [Background] Guice JL, Hollins MD, Farmar JG, Tinker KM, Garvey SM. Microbial inulinase promotes fructan hydrolysis under simulated gastric conditions. Front Nutr. 2023 May 23;10:1129329. doi: 10.3389/fnut.2023.1129329. eCollection 2023. PMID 37305092
- [Background] Van den Houte K, Colomier E, Routhiaux K, Marien Z, Schol J, Van den Bergh J, Vanderstappen J, Pauwels N, Joos A, Arts J, Caenepeel P, De Clerck F, Matthys C, Meulemans A, Jones M, Vanuytsel T, Carbone F, Tack J. Efficacy and Findings of a Blinded Randomized Reintroduction Phase for the Low FODMAP Diet in Irritable Bowel Syndrome. Gastroenterology. 2024 Jul;167(2):333-342. doi: 10.1053/j.gastro.2024.02.008. Epub 2024 Feb 23. PMID 38401741
- [Background] Nagy DU, Sandor-Bajusz KA, Body B, Decsi T, Van Harsselaar J, Theis S, Lohner S. Effect of chicory-derived inulin-type fructans on abundance of Bifidobacterium and on bowel function: a systematic review with meta-analyses. Crit Rev Food Sci Nutr. 2023 Nov;63(33):12018-12035. doi: 10.1080/10408398.2022.2098246. Epub 2022 Jul 14. PMID 35833477